CLINICAL TRIAL: NCT05369780
Title: A Multiple-Dose, Randomized, Double-Blinded, Placebo Controlled Trial To Evaluate The Efficacy Of Hydrolyzed Collagen Peptide On Knees, Hips, and Ankle Pains In Adults With Osteoarthritis
Brief Title: Efficacy Evaluation of Hydrolyzed Collagen Peptide on Knees, Hips, and Ankle Pain in Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sel Sanayi Urunleri Ticaret ve Pazarlama A.S. (Industry)
Collaborators: Alpan Farma Ar-Ge Biyoteknolojileri Ltd.Sti. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ALP-2021-CL-01-2021/01998
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Pain, Joint
MeSH Terms: conditions — Arthralgia | interventions — Collagen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrolized Collagen Peptide (Experimental): This arm will be allocated randomly and receive 10 g hydrolized collagen peptide (Investigational Product) daily throughout the study.
  Interventions: Dietary Supplement: Hydrolyzed Collagen Peptide
- Placebo (Placebo Comparator): This arm will be allocated randomly and receive placebo daily throughout the study.
  Interventions: Dietary Supplement: Hydrolyzed Collagen Peptide

INTERVENTIONS:
Dietary Supplement: Hydrolyzed Collagen Peptide — Dietary Hydrolized Collagen Peptide sourced from bovine
  Other Names: Collagen

SUMMARY:
The aim of this study is to evaluate the effectiveness of Hydrolyzed collagen peptides on joint pain, stiffness and physical function in adults with osteoarthritis who have complaints on knee joints together with hip and ankles. The assessment of improvements on volunteers' quality of life, and safety and tolerability of the product is the other objective of this placebo-controlled, randomized study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female individuals with osteoarthritis on knee who are aged between 45-60 years old,
2. Who are not drug-naïve to osteoarthritis and related conditions,
3. Volunteers who have ability to communicate adequately with the investigator and in agreement to comply with the study requirements,
4. Volunteers who have normal blood pressure and heart rate measured under stabilised conditions at the screening visit after at least 5 minutes of rest under supine position: SBP within 100 to 140 mmHg, DBP within 60 to 90 mmHg and HR within 50 to 100 bpm at least after 5 minutes of rest,
5. Volunteers who have understanding of the study and agreement to give a written informed consent.

Exclusion Criteria:

1. Who have atopic constitution or asthma and/or known allergy for bovine derived collagen products and/or other any of the excipients of the product.
2. Who have hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucosegalactose malabsorption.
3. Who have an active rheumatoid arthritis or any other inflammatory arthritic condition that researchers consider non appropriate.
4. Who have Diabetes Mellitus.
5. Who have the use of oral retinoids or oral steroids in the 6 months prior to initiation of the study.
6. Who have current participation in another clinical study, or participation in a relevant study within 3 months.
7. Who have any history or presence of serious or life-threatening conditions of cardiovascular, neurological, haematological, hepatic, gastrointestinal, renal, pulmonary, endocrinological, metabolism or psychiatric disease, any type of porphiria.
8. Who have the presence or history of malabsorption or any gastrointestinal surgery except appendectomy or except herniotomy.
9. Who are planned to go or already went under a joint-related reconstructive surgery,
10. For female volunteers, who had undergone, or planned to undergo, pregnancy or breastfeeding.
11. Who have current or regular intake of NSAIDS, contraceptives, hormones, obesity drugs, absorption inhibitors or antidepressants
12. Who are suspected to have a high probability of non-compliance to the study procedure and/or completion of the study according to the investigator's judgment.
13. Who have history of drug abuse.
14. Who have relationship to the investigator.
15. Who are not suitable to any of inclusion criteria.
16. Who have history of difficulty of swallowing.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Amelioration on Knee Pain | 2 months
  Amelioration on knee joint pain, stiffness and physical function according to WOMAC (The Western Ontario and McMaster Universities Osteoarthritis Index) score.

SECONDARY OUTCOMES:
Amelioration on Hip Pain | 2 months
  Amelioration on pain, stiffness and physical function of joints of hip according to WOMAC score.
Amelioration on Ankle Pain | 2 months
  Amelioration on pain and physical function of ankles according to AOFASAHFS (American Orthopaedic Foot and Ankle Society Ankle-Hindfoot Scale) scale.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demir-Dora D, Tuna S, Kurtoglu ED, Gursoy S, Balci N, Tezman S, Erenmemisoglu A. Evaluation of the Efficacy and Safety of CollaSel PRO(R) Type I and Type III Hydrolyzed Collagen Peptides in the Treatment of Osteoarthritis: A Double-Blind, Placebo-Controlled, Randomized Clinical Trial. J Clin Med. 2025 May 23;14(11):3655. doi: 10.3390/jcm14113655. PMID 40507417